CLINICAL TRIAL: NCT01464749
Title: Task-oriented Circuit Class Training in Multiple Sclerosis Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, Physical Medicine and Rehabilitation doctor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Multiple Sclerosis TOCT
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; gait rehabilitation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Task-oriented circuit class training (Experimental): Functional Circuit include 6 different work-stations in which patients exercise for 5 minutes in each one : 3 minutes exercises and 2 minutes rest. Total training takes about 30 minutes (2 laps/session over 60 minutes).
  Walking endurance is trained by 30 minutes walking on the treadmill including rests if necessary.
  It is a progressive circuit and subjects, while exercising, receives feedback (visual and auditory) by the physiotherapist. Rests are used to discuss about difficulties and to provide further feedbacks. One task oriented session may include up to 3 patients and lasts 120 minutes. At the end of the 2 weeks an exercises brochure will be given to patients so that they can independently train for 3 month. Independent home training takes about 90 minutes.
  Interventions: Behavioral: Task-oriented circuit class training
- Usual Care (Active Comparator): The control group will not receive any specific rehabilitation treatment for gait performance and mobility improvement (usual care). At any case, the control group will be authorized, at will, to exercise in non-rehabilitative contexts (i.e. swimming, walking, yoga) or do physical rehabilitation in rehabilitative gyms not directly addressed to gait, mobility or balance training such as stretching exercises, active and passive mobilization and Bobath neurorehabilitation or similar.
  Interventions: Behavioral: usual care

INTERVENTIONS:
Behavioral: Task-oriented circuit class training — 5 sessions/week over 2 weeks (10 sessions) 120 minutes/each
  Arms: Task-oriented circuit class training
Behavioral: usual care — no specific rehabilitation
  Arms: Usual Care

SUMMARY:
Aims of the study:

This is a single blind randomized-controlled trial to test the feasibility and the effects of a task oriented training on locomotor function, mobility and balance in multiple sclerosis subjects with moderate gait impairments (EDSS 4 - 5,5). The control group will not be treated with a specific physical therapy (usual care).

Subjects and methods:

60 multiple sclerosis patients will be recruited in an outpatient rehabilitation clinic (Azienda Ospedaliero-Universitaria di Ferrara).

Informed consent will be obtained. Participants will be randomized to (TOCT) task-oriented training (experimental group) or usual care (control group) through a randomization stratification approach, according to a block randomization of 6.

The experimental group will receive 10 task-oriented training sessions over 2 weeks (5 sessions/week=intensive training). Three subjects with a supervisor physiotherapist will take part at the TOCT.

Feasibility outcome will be measured with a specific questionnaire. Treatment efficacy outcome measures will be clinical test for gait speed (10m walking test), walking endurance (six minute walking test), balance (Dynamic Gait Index) and mobility (Time Up and Go Test); a structured interview for the performance(Lower Extremity Mal); self-assessment questionnaire for motor fatigue (Fatigue Severity Scale FSS), multiple sclerosis physical and psychological impact (multiple sclerosis impact scale MSIS-29), walking ability (multiple sclerosis walking scale MSWS-12).

Outcome measures will be assessed the week before the treatment (T0), after the treatment (T1) and at 3 months follow-up (T2) to evaluate treatments retention, by a clinician blinded to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* males and females,
* community dwelling,
* age 18 or older
* diagnosis of multiple sclerosis in a stable phase, with relapses > 3 months prior to study enrollment
* moderate gait impairments referred to Expanded Disability Status Scale (EDSS) between 4 and 5,5

Exclusion Criteria:

* neurologic conditions in addition to multiple sclerosis that may affect motor function
* medical conditions likely to interfere with the ability to safely complete the study
* impaired cognitive functioning: Mini Mental Status Examination < 24

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Feasibility of task-oriented circuit class therapy | 12 months
  It will be performed through the administration of a specific questionnaire

SECONDARY OUTCOMES:
gait speed | 12 months
  10 meter test
mobility | 12 months
  Timed Up and Go
Balance | 12 months
  Dynamic Gait Index
walking endurance | 12 months
  six minute walking test
fatigue | 12 months
  fatigue severity scale
Physical and psychological impact | 12 months
  multiple sclerosis impact scale MSIS-29
Impact on mobility and walking | 12 months
  multiple sclerosis impact scale MSIS-29

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Medicine and Rehabilitation Department Ferrara, Ferrara, Emilia-Romagna, Italy

REFERENCES:
- [Derived] Straudi S, Martinuzzi C, Pavarelli C, Sabbagh Charabati A, Benedetti MG, Foti C, Bonato M, Zancato E, Basaglia N. A task-oriented circuit training in multiple sclerosis: a feasibility study. BMC Neurol. 2014 Jun 7;14:124. doi: 10.1186/1471-2377-14-124. PMID 24906545